CLINICAL TRIAL: NCT01035645
Title: A Single-blind, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of Intravenously Infused GSK1070806 in Healthy and Obese Subjects.
Brief Title: First Time in Human Study of Intravenous Interleukin-18 Antibody
Acronym: A18110040
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110040
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: First time in human; Interleukin-18; Healthy male subjects; Obese male subjects; Monoclonal antibody; Pharmacokinetics; Tolerability; Safety; Pharmacodynamics
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — GSK1070806

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1070806 or placebo (Experimental): This is a single dose escalating study. On enrolment into the study, each subject will be assigned to a group. These groups will be aligned to specific dose levels of GSK1070806. All subjects will be randomised to receive either a single intravenously administered dose of GSK1070806 or matching placebo (saline). The randomisation is generated by GSK prior to study start.
  Interventions: Drug: GSK1070806

INTERVENTIONS:
Drug: GSK1070806 — The study drug, GSK1070806, is a humanised monoclonal antibody. Antibodies are proteins that are made by white blood cells during an immune reaction. They circulate in the blood and attach to foreign proteins called antigens in order to destroy or neutralise them.
  Humanised monoclonal antibodies are a type of protein that is genetically engineered to resemble a human protein (humanised). GSK1070806 is designed to block a specific protein that exists in the body called Interleukin-18. Interleukin-18 works within the immune system, i.e. the body's defence system, which helps protect it from disease, bacteria and viruses. Interleukin-18 activates the immune system to fight infections and may also occasionally cause inflammation.

SUMMARY:
GSK1070806 is a humanised monoclonal antibody that blocks a protein present in the body called Interleukin-18. The main purpose of this study is to test GSK1070806 in healthy and obese male subjects with normal immune systems to find out how safe this drug is and how long the body takes to get rid of it. The study consists of 2 parts. Part 1 will consist of 6 groups of healthy male subjects and Part 2 will consist of 3 groups of obese male subjects. A total of 89 subjects is planned for this study. Subjects in each group will receive one dose of the study drug or placebo. Dosing in Part 2 will not start until dosing of the first 4 groups is completed in Part 1 and the preliminary safety and pharmacokinetic data from these 4 groups in Part 1 has been reviewed. Both parts will be conducted single-blind and with a placebo control. Within each group, allocation of subjects to placebo or active treatment (GSK1070806) will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-65 years inclusive at the time of signing informed consent.
* Subjects must agree to use one of the contraception methods required.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all study assessments.
* Able to read, comprehend and write English at a sufficient level to complete study related materials.
* Healthy as determined by a responsible and experienced physician.
* Positive delayed type hypersensitivity (DTH) reaction to candida antigen within 72 hrs of screening visit (group 4, 8 and 9 subjects only in Part 1).
* Body weight equal or greater than 50kg and BMI within the range of 19-29.9kg/m2 (Part 1 only).
* BMI within the range 30 - 40kg/m2 (Part 2 only).
* Waist circumference >102cm (Part 2 only).
* Fasting plasma insulin >60pmol/L (Part 2 only).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* A positive test for influenza A/B.
* A positive test for Mycobacterium tuberculosis.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units or average daily intake of >3 units. One unit is equivalent to 8 g of alcohol, and the following can be used as a guide: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject is unwilling to abstain from alcohol consumption from 24 hr prior to dosing until discharge from the clinic, and for 24 hr prior to all other out-patient clinic visits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Subject has received live, attenuated or recombinant vaccine(s) within 2 months of randomisation or will require vaccination prior to the time at which plasma levels are predicted to reach an average level of approximately 1.0 µg/mL from when the dose is administered or Day 56 whichever is longer.
* Current evidence, or history within the last 7 days, of an influenza-like illness as defined by fever (>38°C) and two or more of the following symptoms: cough, sore throat, runny nose, sneezing, limb / joint pain, headache, vomiting / diarrhoea in the absence of a known cause, other than influenza.
* Use of anti-Tumor Necrosis Factor (anti-TNF) or anti-Interleukin-1 (anti-IL-1) drugs within 60 days prior to dosing.
* Current evidence of ongoing or acute infection, history of repeated, chronic or opportunistic infections (e.g. recurrent folliculitis, other cutaneous infections or repeated pneumonia) or history of a serious bacterial infection within 6 months of randomisation.
* History of significant cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions that in the opinion of the study physician and/or GSK physician, places the subject at an unacceptable risk as participant in this trial.
* History of Mycobacterium tuberculosis or any other previous Mycobacterium infection.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the study physician and GSK physician the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the study physician or GSK physician contraindicates their participation.
* Current chronic (greater than 3 months) treatment with prescription anti-inflammatory drugs, including corticosteroids and non-steroidal anti-inflammatory drugs.
* History of a severe allergic reaction, angio-edema, anaphylaxis or immunodeficiency.
* History of malignancy, except for adequately treated non-invasive cancer of the skin (basal or squamous cell) (> 2 yrs prior to dosing).
* Subject whose calculated creatinine clearance is less than 80 mL/min
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Subject is unable to refrain from travelling to countries with a high prevalence of infectious disease from when the dose is administered until the time at which the plasma concentration of GSK1070806 is predicted on average to be approximately 1.0µg/mL from when the dose is administered or Day 56 whichever is longer.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Liver function tests above the upper limit of normal at screening (alkaline transaminase (ALT), aspartate transaminase (AST) or bilirubin) (Part 1 subjects only).
* Liver function tests above 2 x the upper limit of normal at screening (alkaline transaminase (ALT), aspartate transaminase (AST)) or 1.5 x the upper limit of normal (bilirubin) (Part 2 subjects only).
* Corrected QT interval (QTc) > 450 msec.
* Subjects who have asthma or a history of asthma, COPD or pneumonia (Note: a subject who suffered from childhood asthma but not as an adult may be included provided they fulfil other entry criteria.)
* Subject has had symptomatic herpes zoster infection within 3 months of randomisation.
* Subjects with a smoking history of >10 cigarettes per day in the last 3 months.
* Experiencing clinically significant ECG abnormalities at screening or at baseline.
* History of elevated blood pressure or current systolic blood pressure > 140mmHg or diastolic blood pressure >90mmHg. (Part 1 only).
* Has a fasting plasma glucose value equal or greater than 7 mmol/L at screening or at baseline, or has been diagnosed with Type 1 or Type 2 diabetes mellitus (Part 2 only)
* Has a fasting triglyceride level >4.52 mmol/L at screening or at baseline. Triglyceride levels within a 5-10% margin above this level will be considered on a case-by-case basis (Part 2 only).
* Subjects currently receiving weight loss treatment such as, but not limited to: "crash"/starvation diets (e.g. <800ckal/day), ALLI™ (Orlistat), Ephedra (ma-huang) or other ephedrine based treatments, Cascara or other herbal treatments which, in the opinion of the investigator and/or GSK Medical Monitor, contraindicates the subject's participation. Subjects must not participate in any of the weight loss treatment outlined above during the course of the study (Part 2 only).
* Subjects planning a substantial change to their diet during the course of the study (Part 2 only).
* Subjects who have participated in a weight loss treatment outlined above within 4 weeks of randomisation (Part 2 only).
* Systolic blood pressure > 150mmHg or diastolic blood pressure > 90mmHg at screening (Part 2 only).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2012-07-11 (Actual); Study Completion 2012-07-11 (Actual)

PRIMARY OUTCOMES:
Adverse events, vital signs, cardiac and ECG parameters and clinical laboratory safety assessments. | From screening upto 56 days for Part 1 subjects in groups 1 and 2. Upto 96 days for group 3 in Part 1 and 126 days for group 4 in Part 1. Upto 56 days for all Part 2 subjects.

SECONDARY OUTCOMES:
Plasma concentrations of GSK1070806 and derived pharmacokinetic parameters thereof. | From dosing upto 56 days for subjects in groups 1 and 2, 152 days for group 3, 213 days for group 4, 274 days for group 8 and upto 300 days in group 9 in Part 1. Upto 152 days for group 5, 213 days for group 6 and 274 days for group 7 subjects in Part 2.
Serum levels of Interleukin-18 (IL-18). | From dosing upto 56 days for subjects in groups 1 and 2, 243 days for group 3, 213 days for group 4, 230 days for group 8 and upto 240 days in group 9 in Part 1. Upto 243 days for group 5, 213 days for group 6 and 230 days for group 7 subjects in Part 2.
Endpoints of immune function and derived pharmacodynamic parameters thereof. | From dosing upto 56 days for subjects in groups 1 and 2, 152 days for groups 3, 8 and 9 and 126 days for group 4 in Part 1. Upto 56 days for all Part 2 subjects.
Serum levels of anti-GSK1070806 binding antibodies. | From dosing upto 56 days for subjects in groups 1 and 2, 243 days for group 3, 213 days for group 4, 274 days for group 8 and 300 days for group 9 in Part 1. Upto 243 days for group 5, 213 days for group 6 and 274 days for group 7 in Part 2.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Mistry P, Reid J, Pouliquen I, McHugh S, Abberley L, DeWall S, Taylor A, Tong X, Rocha Del Cura M, McKie E. Safety, tolerability, pharmacokinetics, and pharmacodynamics of single-dose antiinterleukin- 18 mAb GSK1070806 in healthy and obese subjects. Int J Clin Pharmacol Ther. 2014 Oct;52(10):867-79. doi: 10.5414/CP202087. PMID 25109413
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 110040 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/110040?search=study&search_terms=110040#rs
- Available data/document: Clinical Study Report: 110040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110040 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register